CLINICAL TRIAL: NCT01827241
Title: Outcome of Colonoscopy Screening and Surveillance
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: DR11-0264
Record Dates: First submitted 2013-04-02; First posted 2013-04-09 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Gastroenterology
Keywords: Gastroenterology; Colonoscopy; Screening; Surveillance; Symptom evaluation; Chart review; Data review; Examination findings; Resection techniques; Pathology reports

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Colonoscopy Outcomes: Data collected from endoscopy reports to complete a descriptive analysis of demographics, colonoscopy procedure performance, and assess type of benign colon polyps detected during screening and surveillance from 02/01/2009 - 12/31/2020.
  Interventions: Other: Chart Review

INTERVENTIONS:
Other: Chart Review — Retrospective and prospective data review of colonoscopy procedures, examination findings, resection techniques, and pathology reports.

SUMMARY:
With this study, we plan to review the performance of colonoscopy in colon cancer screening and surveillance, especially with the recent improvements in endoscopic technology (high definition endoscopes), use of split dose preparation which provides excellent colon preparation for detection of lesions and increasing awareness and detection of flat lesions of the colon. The findings will help us define the role of colonoscopy screening of colon polyps and flat lesions and identity areas for improvement. The data will be used for continuing quality improvement and presenting our outcomes at academic meetings and publishing our results in peer reviewed journals.

DETAILED DESCRIPTION:
Investigator's goal is to collect data from the endoscopy reports and clinic station reports to complete a descriptive analysis of the demographics, colonoscopy procedure performance, and assess the type of benign colon polyps detected during screening and surveillance from 02/01/2000 - 12/31/2020.

Specific variable to be reviewed:

1. Patient Demographics: Age, Sex, Race, Height, Weight, BMI (patient privacy will be acknowledged).
2. Indications for Colonoscopy (screening, surveillance, symptoms or tertiary referral [EMR])
3. Comorbid conditions: , cancer and surgical history, medical conditions,
4. Colonoscopy procedure; quality of colon preparation (using the Boston Bowel Preparation Scale) 0 - 3 for each section of the colon (Ascending, Transverse, Descending and Total Colon) , cecal intubation rate, cecal intubation and total procedure time, type of colonoscope (if CO2 was used in the procedure and techniques for colonoscope insertion, including position changes.
5. Examination findings: number of polyps and nature of polyps removed (site, size, surface, vascular pattern); type of polyp removed (serrated and sessile (flat) ; optical features and histology of polyps.
6. Resection techniques: biopsy, snare resection, endoscopic mucosal resection etc.
7. Including Pathology report findings so that a comparison can be made of the optical features and actual pathology report.
8. Outcomes of colonoscopy: adenoma detections (tubular and villous), cancer and quality metrics.
9. Outcome of colonoscopy: Complications (Bleeding and performance).

ELIGIBILITY:
Inclusion Criteria:

1. All Patients who have undergone colonoscopy for screening, surveillance or symptom evaluation.

Exclusion Criteria:

1. None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Chart review from participants receiving colonoscopy at UT MD Anderson Cancer Center in Houston, Texas from 02/01/2009 - 12/31/2020.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2011-09 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Polyp Detection in Colon Cancer Screening and Surveillance | 9 years
  Descriptive tables presented for demographics, polyp counts, colonoscopy experiences, polyp removals and findings. Proportions presented with 95% confidence intervals. Continuous values such as age and times presented with median, minimum and maximum. Comparisons among patient subgroups made with chi-square tests for categorical data and t-tests or the non-parametric alternative, Wilcoxon tests, to compare continuous measures. Graphics such as box plots, trellis plots, bar graphs, or stacked bar graphs used to describe distributions overall and among subgroups.

CONTACTS AND LOCATIONS:
Overall Officials: Gottumukkala S. Raju, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Raju GS, Lum PJ, Ross WA, Thirumurthi S, Miller E, Lynch PM, Lee JH, Bhutani MS, Shafi MA, Weston BR, Pande M, Bresalier RS, Rashid A, Mishra L, Davila ML, Stroehlein JR. Outcome of EMR as an alternative to surgery in patients with complex colon polyps. Gastrointest Endosc. 2016 Aug;84(2):315-25. doi: 10.1016/j.gie.2016.01.067. Epub 2016 Feb 6. PMID 26859866
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org